CLINICAL TRIAL: NCT01469572
Title: Phase IB/II Study of Pasireotide, Everolimus and Selective Internal Radioembolization Therapy (SIRT) for Unresectable Neuroendocrine Hepatic Metastases
Brief Title: Pasireotide, Everolimus and Selective Internal Radioembolization Therapy for Unresectable Hepatic Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Bassel El-Rayes, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00051599; WCI2031-11 (Other: Other)
Record Dates: First submitted 2011-10-13; First posted 2011-11-10 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine hepatic tumors; Liver cancer; Metastatic liver cancer
MeSH Terms: conditions — Neuroendocrine Tumors; Liver Neoplasms | interventions — pasireotide; Sirtuins; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sir-sphere radioembolization (Experimental): Everolimus, Pasireotide and Sir-sphere radioembolization
  Interventions: Drug: Pasireotide; Procedure: Sir-sphere Radioembolization; Drug: Everolimus

INTERVENTIONS:
Drug: Pasireotide — Pasireotide is given as an injection.
  Other Names: SOM230; Signifor
Procedure: Sir-sphere Radioembolization — A catheter will be placed in a branch of the hepatic artery (liver) that supplies the tumor with blood. Radioactive beads will be injected into the tumor through the catheter.
  Other Names: Selective Internal Radioembolization Therapy; SIRT
Drug: Everolimus — Given orally every day for the duration of the study
  Other Names: RAD001; Afinitor

SUMMARY:
The purpose of this study is to see the safety and activity of using pasireotide, everolimus and radioembolization (Selective Internal Radioembolization Therapy-SIRT) in the treatment of neuroendocrine tumors (carcinoid) that has spread to the liver. Both everolimus or radioembolization are considered "standard of care" regimens in patients with liver lesions from neuroendocrine tumors. However, the use of the combination of everolimus and radioembolization has not been formally evaluated in the setting of a clinical trial. Pasireotide is a medication that is intended to block the hormonal secretions from the neuroendocrine tumors.

This study is divided into two parts. In the first part, the aim of the study is to determine the safety of combining everolimus, pasireotide, and radioembolization. For this part of the study the investigators will enroll up to 18 patients. After the investigators confirm the safety of the combination, they will conduct the second part of the study which will focus on evaluating the effectiveness of the combination. For this part of the study the investigators intend to enroll a total of 37 patients.

DETAILED DESCRIPTION:
Liver metastasis remain a major challenge in the care of patients with Neuroendocrine Tumors (NET). This study is evaluating the combination of systemic therapies plus radioembolization for the treatment of liver metastasis from NET. The study allows pancreatic and intestinal NET that have spread to the liver.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed low to intermediate grade neuroendocrine tumors with unresectable liver metastasis
2. Patients must have evidence of disease progression by Response Evaluation Criteria in Solid Tumors (RECIST) despite optimal octreotide therapy (octreotide long acting release [LAR] 30 mg every month)
3. Prior treatment permitted include: surgery, prior systemic therapies (≤ 2 prior lines of chemotherapy), or radiation therapy
4. Patients must have measurable disease by RECIST 1.1 criteria
5. For the patients in the phase Ib study, neuroendocrine tumor must involve both liver lobes
6. Minimum of four weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy (adequately recovered from the acute toxicities of any prior therapy)
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
8. Adequate bone marrow function as shown by:

   * Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L
   * Platelets greater than or equal to 100 x 10^9/L
   * Hb greater than 9 g/dL
9. Adequate liver function as shown by:

   * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5x ULN (≤ 3x ULN in patients with liver metastases)
10. International normalized ratio (INR) ≤ 1.5 (anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin)
11. Patient receiving low molecular weight (LMW) heparin on stable therapeutic dose for more than 2 weeks or with factor Xa level < 1.1 U/mL can be enrolled if LMW heparin can be safely discontinued at least 24 hours prior to invasive vascular procedures (angiography and SIR-sphere administration)
12. Adequate renal function: serum creatinine ≤ 1.5 x ULN
13. Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
14. Women of childbearing potential must have a negative serum pregnancy test within 14 days of the administration of the first study treatment. Women must not be lactating. Both men and women of childbearing potential must be advised of the importance of using effective birth control measures during the course of the study.
15. Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator (or his/her designee) with the aid of written information.

Exclusion Criteria:

1. Evidence of ascites, cirrhosis, portal hypertension or portal vein thrombosis
2. Prior radiation to the upper abdomen
3. Contraindications to angiography
4. Patients with extensive tumor replacement of the liver defined as tumor volume > 50% of liver
5. Lung shunt ≥ 20%
6. Prior treatment with any investigational drug within the preceding 4 weeks
7. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
8. Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, bacillus Calmette-Guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines.
9. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
10. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
11. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

    * Symptomatic congestive heart failure of New York Heart Association Class III or IV
    * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
    * Severely impaired lung function as defined as spirometry and diffusing capacity of lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
    * Uncontrolled diabetes as defined by hemoglobin A1C (HbA1c) > 7% despite therapy.
    * Active (acute or chronic) or uncontrolled severe infections
    * Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C)
12. History of liver disease such as cirrhosis or chronic active hepatitis. Presence of Hepatitis B surface antigen (HepBSAg) or presence of hepatitis C antibody. History of, or current alcohol misuse/abuse within the past 12 months
13. Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result (ELISA and Western blot)
14. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
15. Patients with an active, bleeding diathesis
16. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug, by both sexes. (Women of childbearing potential [WOCBP] must have a negative urine or serum pregnancy test within 14 days prior to administration of pasireotide and everolimus) Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
17. Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
18. Patients who have received prior treatment with an mammalian target of rapamycin (mTOR) inhibitor (e.g., sirolimus, temsirolimus, everolimus).
19. Patients with a known hypersensitivity to everolimus or other rapamycins (e.g., sirolimus, temsirolimus) or to its excipients
20. Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR formulations
21. History of noncompliance to medical regimens
22. Patients unwilling to or unable to comply with the protocol
23. QT related exclusion criteria include:

    * QT Fridericia's Correction Formula (QTcF) at screening > 450 msec
    * History of syncope or family history of idiopathic sudden death
    * Sustained or clinically significant cardiac arrhythmias
    * Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade atrioventricular (AV) block
    * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
    * Concomitant medication(s) known to increase the QT interval
24. Known gallbladder or bile duct disease, acute or chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-12; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the number of patients who develop side effects from combination therapy. | 1 month
  Determine the maximum tolerated dose of pasireotide and everolimus that can be administered with SIR spheres. Patients will be treated in cohorts of three. Dose of everolimus will be increased after every three patients. Plan is to determine the maximum dose that can be administered with less than 2 out of 6 patients develop significant side effects.

SECONDARY OUTCOMES:
Compare the size of the tumor before and three months after treatment using cross sectional imaging (CT ro MRI) | 3 months
  To evaluate the response rate associated with the combination of pasireotide, everolimus and radioembolization. Response is defined as radiologic shrinkage in the size of the tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Bassel El-Rayes, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Kim HS, Shaib WL, Zhang C, Nagaraju GP, Wu C, Alese OB, Chen Z, Brutcher E, Renfroe M, El-Rayes BF. Phase 1b study of pasireotide, everolimus, and selective internal radioembolization therapy for unresectable neuroendocrine tumors with hepatic metastases. Cancer. 2018 May 1;124(9):1992-2000. doi: 10.1002/cncr.31192. Epub 2018 Feb 16. PMID 29451701